CLINICAL TRIAL: NCT00484926
Title: Correlation of Clopidogrel Therapy Discontinuation in REAL-world Patients Treated With Drug-Eluting Stent Implantation and Late Coronary Arterial Thrombotic Events
Brief Title: Association of Clopidogrel Therapy and Stent Thrombosis
Acronym: REAL-LATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20070186
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Coronary Artery Disease
Keywords: coronary disease; stents; antiplatelet drugs; drug-eluting stents
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Active Comparator): Aspirin monotherapy (stopping clopidogrel at 1 year after DES)
  Interventions: Drug: Aspirin monotherapy
- Aspirin,Clopidogrel (Experimental): Aspirin,Clopidogrel Dual antiplatelet therapy (continue aspirin and clopidogrel 1year after DES)
  Interventions: Drug: Aspirin,Clopidogrel

INTERVENTIONS:
Drug: Aspirin monotherapy — stopping clopidogrel at 1 year after DES
  Arms: Aspirin
Drug: Aspirin,Clopidogrel — continue aspirin and clopidogrel 1year after DES
  Other Names: Aspirin,Clopidogrel Dual antiplatelet therapy
  Arms: Aspirin,Clopidogrel

SUMMARY:
The purpose of REAL-LATE (Correlation of Clopidogrel Therapy Discontinuation in REAL-world Patients Treated with Drug-Eluting Stent Implantation and Late Coronary Arterial Thrombotic Events) trial is to assess the relationship between clopidogrel use and long-term rates of cardiac death or MI after DES implantation in real-world practice and to estimate the duration of dual antiplatelet therapy for preventing the late thrombotic events.

DETAILED DESCRIPTION:
An observational analysis from BASKET-LATE (Basel Stent Kosten-Effekivitats Trial-Late Thrombotic Events) examined the incidence of clinical events after cessation of clopidogrel therapy. This study identified 746 patients who were without major adverse events 6 months after drug-eluting or bare-metal stent placement. All patients had stopped taking clopidogrel and were followed up for an additional 12 months. At 18-month follow-up, there was no difference between patients with a drug-eluting or bare-metal stent in cumulative rates of death or myocardial infarction (MI). However, after clopidogrel discontinuation patients receiving drug-eluting vs bare-metal stents experienced higher rates of death and MI (4.9% vs 1.3%, respectively). These results have created uncertainty regarding the minimal necessary duration of antiplatelet therapy after drug-eluting stent implantation. Also, there remains widespread uncertainty regarding the risk of clinical events after the discontinuation of clopidogrel, particularly after DES implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Among consecutive patients treated with DES, event-free patients who survived at least the first 12 months without nonfatal MI or repeat revascularization
2. The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

1. Contraindication to antiplatelet therapy (aspirin or clopidogrel)
2. Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
3. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
4. Concurrent bleeding diathesis or major bleeding history requiring discontinuation of antiplatelet drugs.
5. Patients with left main stem stenosis (>50% by visual estimate) or left main stenting
6. Concomitant disease requiring long-term use of clopidogrel (stroke, peripheral vascular disease, significant carotid a. disease, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2007-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The composite of cardiac death or MI in the intent-to-treat population | 1 year after randomization

SECONDARY OUTCOMES:
All death | 1 year after randomization
Myocardial infarction | 1 year after randomization
Stroke | 1 year after randomization
Stent Thrombosis | 1 year after randomization
Bleeding events | 1 year after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Department of Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (13):
- South Korea (13):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Choeng Ju St.Mary's Hospital, Choeng Ju
  - Kangwon National University Hospital, Chuncheon
  - Chungnam National University Hospital, Daejeon
  - Asan Medical Center, Gangneung
  - DongGuk University Gyongju Hospital, Gyongju
  - Chonbuk National University Hospital, Jeonju
  - Kwangju Christian Hospital, Kwangju
  - Asan Medical Center, Seoul
  - Hangang Sacred Heart Hospital, Seoul
  - Kyungsang University Hospital, Seoul
  - Seoul Veterans Hospital, Seoul
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Derived] Park SJ, Park DW, Kim YH, Kang SJ, Lee SW, Lee CW, Han KH, Park SW, Yun SC, Lee SG, Rha SW, Seong IW, Jeong MH, Hur SH, Lee NH, Yoon J, Yang JY, Lee BK, Choi YJ, Chung WS, Lim DS, Cheong SS, Kim KS, Chae JK, Nah DY, Jeon DS, Seung KB, Jang JS, Park HS, Lee K. Duration of dual antiplatelet therapy after implantation of drug-eluting stents. N Engl J Med. 2010 Apr 15;362(15):1374-82. doi: 10.1056/NEJMoa1001266. Epub 2010 Mar 15. PMID 20231231